CLINICAL TRIAL: NCT04715139
Title: A Multi-Center, Prospective Registry to Evaluate the Continued Safety and Performance of the Foot and Ankle Products
Brief Title: Evaluate the Continued Safety and Performance of the Foot and Ankle Products
Status: Recruiting | Type: Observational
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AIRR-0006
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-06

CONDITIONS: Hyperpronated Foot; Reconstruction Surgeries of the Foot; Fixation of Fractures and Fusion (Bunionectomy Osteotomies) of the Foot/Ankle; Fixation of Small Bone Fragments of the Foot/Ankle; Lisfranc Arthrodesis; Mono or Bi-cortical Osteotomies in the Forefoot; First Metatarsophalangeal Arthrodesis; Akin Osteotomy; Midfoot and Hindfoot Arthrodeses or Osteotomies; Fixation of Osteotomies for Hallux Valgus Treatment (Scarf and Chevron); Arthrodesis of the Metatarsocuneiform Joint to Reposition and Stabilize Metatarsus Primus Varus; Osteotomy Fixation of Hallux Valgus Repair (Such as Scarf and Chevron Etc.); Medial Ankle Stabilization; Tibiotalocalcaneal Arthrodesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Products listed in Descriptions: * ProStop
  * BioCompression Screw
  * TRIM-IT Drill Pin/TRIM-IT Spin Pin
  * Headless Compression Screw/Compression FT Screw
  * DynaNite Nitinol Staple
  * BioComposite SutureTak Anchor
  * Beveled Headed FT Screw
  * KreuLock Screws
  * ArthroFLEX dermal allograft
  * DualCompression Hindfoot Nail
  Interventions: Device: Products listed in Group/Cohort Description

INTERVENTIONS:
Device: Products listed in Group/Cohort Description — Depending on approved indication per product

SUMMARY:
The objective of the registry is to evaluate the continued safety and performance of Arthrex foot and ankle products, including the ProStop® implant for hyperpronated foot; Bio-Compression Screw for reconstruction surgeries of the foot; TRIM-IT Drill Pin® system and/or TRIM-IT Spin Pin™ system for fixation of fractures and fusion (bunionectomy osteotomies) of the foot/ankle; Headless Compression Screws and Compression FT Screws for fixation of small bone fragments of the foot/ankle; DynaNite® nitinol staple for midfoot and hindfoot arthrodeses or osteotomies, first metatarsophalangeal arthrodesis, and mono or bi-cortical osteotomies in the forefoot; BioComposite SutureTak® anchor for medial ankle stabilization; Beveled FT Screws for hallux valgus repair; KreuLock™ screws for ankle fractures; ArthroFLEX® dermal allograft for hallux rigidus arthroplasty; and DualCompression Hindfoot Nail for tibiotalocalcaneal arthrodesis.

DETAILED DESCRIPTION:
Device-related adverse events will be continuously assessed and summarized at three months, six months, one year, and two years postoperatively to evaluate safety. A physical exam of the target area will be conducted three months postoperatively to evaluate performance. Range of motion (ROM) will be assessed preoperatively, at three months, six months, and one year postoperatively for the ArthroFLEX® dermal allograft only. Patient-reported outcomes (PROs) will be evaluated for all products at three months, six months, and one year. Additionally, PROs will be assessed at two years postoperatively for ArthroFLEX® dermal allograft and DualCompression Hindfoot Nail only. PROs include the Foot and Ankle Ability Measures (FAAM), Visual Analogue Scale (VAS), Single Assessment Numeric Evaluation (SANE) score, and Veterans Rand 12-Item Health Survey (VR-12). DualCompression X-rays will be evaluated at six months and one year postoperatively for ArthroFLEX® dermal allograft and DualCompression Hindfoot Nail only, and CT scans will be assessed at three months postoperatively for DualCompression Hindfoot Nail only.

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires surgery using Arthrex foot and ankle products included in the registry.
2. Subject is 18 years of age or over (all products except ProStop®).
3. Subject age >two to 17 years (ProStop® product only).
4. Capable of completing self-administered questionnaires.
5. Willing and able to return for all study-related follow-up visits.
6. Subject or subject's representative signed informed consent and assent, when applicable, and is willing and able to comply with all study requirements.

   (ArthroFLEX® subjects only):
7. Degenerative or post-traumatic arthritis of the 1st MTP joint with grade 2, 3, or 4.
8. Subjects who require surgical intervention or are medically indicated for an arthrodesis or arthroplasty of the 1st MTP.

   DualCompression Hindfoot Nail subjects only:
9. The participant must have instability, arthritis, rigid deformity, or severe foot or ankle deformity necessitating tibiotalocalcaneal arthrodesis, commonly referred to as TTC arthrodesis.
10. The participant should be undergoing treatment with the Arthrex DualCompression Hindfoot Nail, either as a primary procedure or as a revision surgery, per standard of care

Exclusion Criteria:

1. Insufficient quantity or quality of bone.
2. Blood supply limitations and previous infections, which may retard healing.
3. Foreign-body sensitivity.
4. Any active infection or blood supply limitations.
5. Conditions that tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period.
6. Subjects that are skeletally immature (except for ProStop®).
7. Subject is considered from vulnerable population (i.e., child, prisoner, pregnant).
8. Subjects who are contraindicated for these devices.
9. Subject is currently receiving compensation or benefits due to a work-related injury or illness under any applicable occupational injury or disability program.
10. Subject has a planned or scheduled additional surgery on the affected or contralateral lower extremity within the course of the study.

    (® Nitinol Staple Subjects only):
11. Subjects who have a comminuted bone surface that would not allow for staple placement as required by the DynaNite® Nitinol Staples directions for use.
12. Subjects who have pathologic bone conditions such as osteopenia that would impair the ability to securely fix the implant as required by the DynaNite® Nitinol Staples directions for use.

    (ArthroFLEX® subjects only):
13. Additional ipsilateral lower limb pathology that requires active treatment.
14. Bilateral degenerative or post-traumatic arthritis of the 1st MTP joints that would require simultaneous treatment of both MTP joints.
15. Diagnosis of gout.
16. Any significant bone loss, avascular necrosis, and/or large osteochondral cyst (>1cm) of the 1st MTP joint.
17. Lesions greater than 10mm in size.
18. Hallux varus to any degree, or hallux valgus >20 degrees.

    (DualCompression Hindfoot Nail subjects only):
19. Requiring only a tibiotalar or subtalar arthrodesis
20. Patient requires bulk allograft or metal spacer implant to fill large bony defect and aid in limb salvage

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 700 subjects (50 subjects per product/indication pair) will be enrolled. The subject population will be male and female,18 years of age or older, with the exception of ProStop®, which includes subjects aged >2 to 17 years of age. Subjects will be recruited from the surgeon's patient population or referrals from other physicians.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess change in Visual Analogue Scale (VAS) survey | preoperatively, 3 months, 6 months and 12 months post operative
  Patient reported pain scale 0-10 point scale (0 min, 10 max)
To assess changes in Veterans RAND Health (VR-12) survey | preoperatively, 3 months, 6 months and 12 months post operative
  Patient reported changes in general health and mental survey. Average score is 50 (negative answers bring scores down, positive answers bring score up)
To assess changes in Foot and Ankle Ability Measures (FAAM) survey | preoperatively, 3 months, 6 months and 12 months post operative
  Patient reported change to physical function for individuals with foot and ankle related impairments. A higher score represents a higher level of physical function
To assess change in Single Assessment Numeric Evaluation (SANE) survey | preoperatively, 3 months, 6 months and 12 months post operative
  Patient reported change to affected body part on a scale from 0 to 100, with 100 representing their normal function.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - UC Davis Medical Center, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - TOA Research Foundation, Nashville, Tennessee
  - Barrett Podiatry, San Antonio, Texas
  - Atlantic Orthopaedic Specialists, Virginia Beach, Virginia
- OrthoPedes, Duisburg, Germany
- Dr Haroun Mahomed Orthopaedic Practice, Durban, South Africa

IPD SHARING:
Plan to Share IPD: Undecided